CLINICAL TRIAL: NCT06800599
Title: Registro Mono-istituzionale Di Individui Sottoposti a Valutazione Del Rischio Genetico Oncologico
Brief Title: Single-institution Register of Individuals Undergoing Cancer Genetic Risk Assessment
Status: Enrolling by invitation | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Other Study IDs: REGIO
Record Dates: First submitted 2024-11-28; First posted 2025-01-30 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2024-10

CONDITIONS: Genetic Predisposition to Cancer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 15 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Prospective: During oncology genetic counselling, together with the standard forms usually applied, the information sheet concerning participation in the register will also be sent to users who meet the inclusion criteria.
- Retrospective: For patients who underwent oncological genetic counselling before the start of the registry, retrospective recruitment will be carried out by means of re-contact for the purpose of proposing joining the registry.

SUMMARY:
Single-centre, retrospective, prospective observational cohort study, based on the registration of data from users of the Oncology Genetics Outpatient Clinic

DETAILED DESCRIPTION:
The primary objective of this study is to establish a register to collect and update over time the clinical, genetic and socio-demographic data of all patients who will be assessed for a suspected oncological genetic predisposition, in order to acquire information that can be used for conducting specific studies aimed at clarifying the various uncertainties that still characterise these diseases, such as the clinical significance and the genotype-phenotype correlations of many alterations in oncological predisposition genes oncological predisposition genes, the clinical and bio-pathological features predictive of a significant probability of identifying mutations in these genes, the efficacy of surveillance and prevention measures undertaken to reduce the risk oncological risk according to guidelines, the effectiveness of oncological therapies in patients with hereditary tumours in comparison with those with sporadic neoplasms sporadic neoplasms, risk perception, emotional impact and also interpersonal experiences associated with oncological genetic risk assessment.

These are objectives of primary interest to both the patient and public health (given the general frequency of oncological diseases), because the information acquired will make it possible to improve the general clinical management of all cancer patients and their families.

ELIGIBILITY:
Inclusion Criteria:

* participants aged 0 days or older at the time of genetic counselling
* obtaining a signed informed consent

Exclusion Criteria:

* misdiagnosis of oncological counselling during oncological genetic counselling

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All users attending Oncology Genetics outpatient clinics will be registered. The user population of these outpatient clinics includes all patients assessed for hereditary cancer risk regardless of age, gender, disease status and genetic testing. The register will include both the proband, i.e. the first person in the family to undergo an oncological genetic assessment, and any family members who perform the assessment subsequently.
Sampling Method: Non-Probability Sample
Enrollment: 7000 (Estimated)
Dates: Start 2022-05-01 (Actual); Primary Completion 2037-12-31 (Estimated); Study Completion 2037-12-31 (Estimated)

PRIMARY OUTCOMES:
Register and follow up over time individuals assessed for suspected genetic predisposition to cancer | 15 years
  Register and follow up over time individuals assessed for suspected genetic predisposition to cancer

SECONDARY OUTCOMES:
Possibility of conducting studies targeted at specific objectives | 15 years
  Acquire information that can be used for conducting specific studies aimed at clarifying the various uncertainties that still characterize these cancer diseases due to genetic predisposition

CONTACTS AND LOCATIONS:
Overall Officials: Daniela Turchetti, MD, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna, Policlinico di Sant'Orsola
Locations (1):
- IRCCS Azienda Ospedaliero-Universitaria di Bologna, Policlinico di Sant'Orsola, Bologna, Italy, Italy

IPD SHARING:
Plan to Share IPD: No